CLINICAL TRIAL: NCT05235399
Title: Exploring Right vEntricular Function Applicability in a Prediction mOdel to Identify pReterm infanTs With Early BronchoPulmonary Dysplasia (REPORT - BPD Study): a Mixed Methods Observational Cohort Feasibility Study
Brief Title: Right vEntricular Function Prediction mOdel to Identify pReterm infanTs With Early BronchoPulmonary Dysplasia.
Acronym: REPORT-BPD
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: 22/NEO/636; 311906 (Other: IRAS)
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-01

CONDITIONS: Bronchopulmonary Dysplasia; Right Ventricular Dysfunction; In the Perinatal Period
Keywords: Right ventricular function; Bronchopulmonary Dysplasia; Prematurity; Neonates; Echocardiography
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Ventricular Dysfunction, Right; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants who are born before 32 weeks of gestation.: The study aims to recruit preterm infants who are born before 32 weeks of gestation.
  Interventions: Other: Echo scans

INTERVENTIONS:
Other: Echo scans — Echo heart scan will be performed on the participating preterm infants on the 5th and 9th day of postnatal life.

SUMMARY:
Short title REPORT-BPD feasibility study

Design A mixed methods observational cohort feasibility study

Study Setting Neonatal Intensive Care Unit at University Hospitals Plymouth NHS Trust

Aim To explore the feasibility of measuring the right ventricular function of the premature heart to develop a prediction model to identify early BronchoPulmonary Dysplasia in premature infants.

Objectives 1. To assess the feasibility and acceptability of the study procedures e.g., recruitment, echo scans performance, data collection, storage, and analysis.

2. To identify the sensitive echo parameters in assessing the right ventricle function of the heart to be included in a prediction model to identify early BPD in premature infants.

Study Participants Preterm infants born <32 weeks of gestational age, their parents and healthcare professionals involved in the care of the study's preterm infants.

Sample size 40 preterm infants

Follow-up Each preterm infant will be followed up till they are 36 weeks of post menstrual age (PMA) or until discharge home whichever comes first.

Study Period 18 months

Outcome Measures

1. Establishing sensitive and feasible echo parameters for detecting right ventricle dysfunction associated with early BPD pulmonary vascular changes.
2. Suitability of eligibility criteria and sample characteristics.
3. Fidelity to the study procedures such as recruitment, data collection including echo scans performance at the set time points.
4. Recruitment, accrual, and retention rates.

DETAILED DESCRIPTION:
RATIONALE The current research findings demonstrated a persistently elevated myocardial performance index of the right ventricle (RV) in the first two weeks of postnatal life (WoPL) in preterm infants with incipient BPD. The identification of the early myocardial dysfunction of RV that is associated with early pulmonary vascular disease (PVD) through echo scan examination in the first two WoPL can potentially serve as a marker for detecting preterm infants with an early BPD.

Data from 1,735 infants born between 23-30 weeks of gestational age (GA) showed that the proportion of preterm infants born < 31 weeks needing oxygen decreases from birth to the 7th day of postnatal life (DoPL). This is followed by a steep rise in the number of infants requiring oxygen in the same cohort at the start of the second week of postnatal life (WoPL). The number of preterm infants needing extra oxygen, peaks at the 14th DoPL. These studies indicate that the pathological pulmonary changes start as early as the first 10 DoPL. Furthermore, studies have identified the end of the first week of postnatal life (WoPL) and the beginning of the second WoPL as the time point when early respiratory problems start to surface. According to the vascular theory, the pathological processes affecting the pulmonary vascular bed are already happening before the appearance of the clinical signs associated with early BPD. The proposed study (REPORT-BPD) aims to capture the early burden exerted on the RV by early BPD and its associated pulmonary vascular changes through performing functional echo examinations at two time points, 5th and 9th day of postnatal life (DoPL) and utilising the findings to construct a prediction model.

To our knowledge, no study has used functional echo examinations to assess extra load or strain imposed by early BPD on the RV on the two time points (5th & 9th DoPL) in the first 10 DoPL.

The cardiac muscle of the preterm infant's heart has premature function. The premature heart reduced contractility is secondary to several reasons such as less myofibrils per cross-sectional area together with immature internal organisation. In addition, there is a lower number of β-adrenergic receptors and underdeveloped sympathetic nervous network. Furthermore, the underdeveloped intrinsic myocardial function following preterm birth is the result of abnormal right ventricle performance with remodelling after birth that persists in the first year of life.

Current research supports the vascular theory as the main pathophysiology of BPD i.e., the pathological process of BPD starts in the pulmonary vascular bed prior to the involvement of the parenchyma of the lungs. So, when the early BPD respiratory insufficiency starts to manifest clinically on 7th day of postnatal life, the adverse haemodynamic changes are already ongoing. In addition, the immaturity of the right ventricle (RV) will render the RV more sensitive to the extra burden imposed by the negative haemodynamic effects of early BPD causing worsening of the RV dysfunction.

In summary, the rationale of the study is outlined nicely by a quote from Niccolo Michiavelli; an Italian diplomat, philosopher and historian, who lived during the renaissance (1469 - 1527):

"In the beginning of the malady it is easy to cure but difficult to detect, but in the course of time, not having been either detected or treated in the beginning, it becomes easy to detect but difficult to cure." To the best our knowledge, this is the first study that assesses the right ventricle dysfunction through two echo scans performed at two specified time points before and after the 7th day of postnatal life when early BPD respiratory insufficiency starts to be evident. Then, the data generated will be utilised to formulate a prediction model for early BPD. In other words, since it is very difficult to diagnose early BPD, this study will utilise highly specialised technologies in analysing the echo images and the data generated will be used to formulate a prediction model to identify BPD at its early stage. Additionally, the rationale behind incorporating qualitative work is because it is important to explore the experiences of parents and clinicians in participating in REPORT-BPD study to inform the design of a larger trial by addressing any gaps identified during this study.

OBJECTIVES

1. To assess the feasibility and acceptability of the study procedures e.g., recruitment, echo scans performance, data collection, storage, and analysis.
2. To identify the sensitive echo parameters in assessing the right ventricle function of the heart to be included in a prediction model to identify early BPD in premature infants.

STUDY DESIGN This is a longitudinal, observational, cohort and feasibility study. STUDY SETTING This study will be conducted at the regional tertiary neonatal intensive care unit (NICU) at University Hospitals Plymouth NHS Trust (UHP), Plymouth. The total NICU capacity is 40 neonatal admissions (6 intensive care cots, 6 high dependency care cots, 10 special care cots and 18 cots in transitional care ward).

SAMPLE AND RECRUITMENT

Sample size

The exploratory nature of this feasibility study dictated to set a realistic target of recruiting 40 preterm infants who are born before 32 weeks of gestation.

The regional tertiary NICU at the UHP admitted 89, 101 and 69 preterm infants who were born before 32 PMA in the years 2018, 2019 and 2020, respectively. Based on the careful examination of the data of the admissions in 2018; two thirds of these preterm infants met the inclusion criteria of the proposed study with one third of them i.e., eligible preterm infants developed moderate - severe BPD.

Therefore, the proposed feasibility study realistic sample size is 40 preterm infants over an 18-month recruitment period.

Participants

The participant whose data will be subjected to the trial analysis - both for the primary analysis and any applicable secondary analyses are:

1. Infants survived till the gestational age when the diagnosis of no BPD or BPD with its severity can be established.
2. Infants who died before the set gestational age (36 weeks PMA) with severe BPD is being the main cause of death.

   Participant identification

   The identification of eligible infants for the study will be carried out by the neonatal clinical team once a preterm infant is admitted to the regional tertiary NICU at UHP, either from the delivery suite in UHP or from another neonatal unit in the region for continuity of care. The neonatal clinical team will be consisted of the clinicians who are working in the neonatal unit such as, consultant neonatologists, trainee doctors, advanced neonatal nurse practitioners, neonatal staff nurses. While the neonatal research team is consisted of the clinicians such as, consultant neonatologists, trainee doctors and advanced nurse practitioners, who are good clinical practice (GCP) trained and registered in the study delegates' log.

   The neonatal clinical team will inform the neonatal research team of the potential recruits to instigate the recruitment process.

   Screening

   The screening process will occur on the possible two time points:
   * Timepoint 1: If possible, antenatal screening will be carried out. The obstetric or midwifery team will inform the neonatal clinical team of the admitted women with preterm labour. This will be followed by screening for eligibility by the clinical neonatal team by reviewing the medical notes. Then the clinical neonatal team will inform the neonatal research team if the unborn infant is deemed a potential recruit so the initial conversation can happen antenatally.
   * Timepoint 2: If screening is not possible at timepoint 1 parents of the suitable preterm infants will be approached in the second day after the birth of their infant.

   A screening log will be maintained.

   Consent

   All parents will be spoken to in person by the neonatal research team, who are also part of the neonatal clinical team, in the antenatal wards, in the delivery suite antenatally or in the neonatal unit postnatally. The neonatal research team members will clearly introduce themselves and state that this conversation will be about the parents and their preterm infants' participation in REPORT-BPD study. The talk will focus on providing a clear verbal explanation of the research project and why the parents and their preterm infants are invited to participate in this study, together with giving them a patient/parent information sheet (PIS) and informed consent form. The parents will also be given contact details for the chief investigator (CI) and the neonatal research team in case they wish to seek further information about the study.

   Informed and written consent to enter the study will be sought from each participant, in this case participants' parents. Signed parents' informed consent forms will be obtained prior to the participation in the study. If parents are interested in participating, a neonatal consultant, a senior trainee doctor or senior advanced nurse practitioner who is a member of the neonatal research team, will be able to dedicate some of their time to obtain consent at the second day after the birth of the potential recruit. All participants will be made aware that they are free to withdraw at any time from the study without giving reasons and without prejudicing further treatment.

   A delegation log will be maintained to ensure that the medical practitioners registered as a study delegate who are participating in the consenting process of this study, are duly authorised, completed a Good Clinical Practice (GCP) training, experienced clinicians and competent to participate according to the ethically approved protocol, principles of GCP and Declaration of Helsinki.

   DATA COLLECTION

   As per the standards of care echo scans are performed when one or more of the following clinical indications are present:
   * Preterm infants who require mechanical ventilation or non-invasive respiratory support (CPAP ≥ 4 cm H2O, High Flow ≥ 4 L/min).
   * Detection of a cardiac murmur in the first three days after birth.
   * Assessment of patent ductus arteriosus (PDA).
   * Preterm infants have central line in-situ, so echo is needed to assess line position.

   Three Data Collection Time Points

   Data Collection Point 1: First echo scan will be performed on the 5th Day of postnatal life (DoPL) together with the following data will be collected:
   * Current weight in grams.
   * Vital signs:

     o Heart rate.

     o Respiratory rate.

     o Oxygen saturation.
     * Temperature.
     * BP including systolic, diastolic, and mean BP.
   * Acquisition of the echo scan images.
   * Ventilatory support:

     o Mode of ventilation.

     o Mean airway pressure (MAP) used.

     o FiO2.

     2) Second echo scan will be performed on the 9th DoPL with the following will be collected:
   * Infant's weight in grams.
   * Vital signs:

     o Heart rate.

     o Respiratory rate.
     * Oxygen saturation.
     * Temperature.
     * BP including systolic, diastolic, and mean BP.
   * Acquisition of the echo scan images.
   * Ventilatory support:

     o Mode of ventilation.

     o Mean airway pressure (MAP) used.

     o FiO2.

     3) At 36 weeks of PMA or at discharge if discharged home before 36 weeks of PMA:
   * Ventilatory support:

     * Mode of ventilation.
     * Mean airway pressure (MAP) used.
     * FiO2.
   * Outcomes.

   STATISTICS AND DATA ANALYSIS

   The distribution of all continuous variables will be visualised to check for normality and summarised using appropriate descriptive statistics. At 36 weeks, infants will be categorised into two groups: (i) moderate or severe BPD and (ii) mild or no BPD.

   In order to help identify potential candidate variables for inclusion in a predictive model the following analyses will be undertaken. Differences in clinical characteristics and echo scan parameters between the two groups of infants will be visualised using boxplots. The comparison between the two groups will be further assessed using t-tests for normally distributed continuous variables and Mann-Whitney U tests for non-normally distributed variables. Chi-squared tests will be used to compare categorical variables between groups.

   The association among clinical and echo parameters will also be explored through visualisation using scatterplots and Pearson's or Spearman's correlations as appropriate. Analyses will be considered exploratory in nature and as such no adjustment for multiple comparisons will be made - interpretation of these analyses will consider the estimates of the between group differences and their 95% confidence intervals. Comparative analyses of the changes between the two timepoints when the echo scans performed i.e., 5th and 9th day of postnatal life, will be conducted.

ELIGIBILITY:
INCLUSION CRITERIA

* Born at < 32 weeks gestational age.
* The echo scans are indicated as per the recommended neonatal practice:

  * Preterm infants who require mechanical ventilation or non-invasive respiratory support (CPAP ≥ 4 cm H2O, High Flow ≥ 4 L/min).
  * Detection of a cardiac murmur in the first three days after birth.
  * Assessment of patent ductus arteriosus (PDA).
  * Preterm infants have central line in-situ, so echo is needed to assess line position.

EXCLUSION CRITERIA

* Preterm infants with major congenital anomalies, such as pulmonary hypoplasia or congenital heart disease (except PFO or PDA).
* Preterm infants with a poor prospect of survival.
* Preterm infants whose parents do not consent.
* Preterm infants who are still in need of blood pressure supporting medications, such as, (inotropes) when the study echo scans are due.
* Preterm infants need inhaled nitric oxide gas when the study echo scans are due.

PDA - patent ductus arteriosus, PFO - patent foramen ovale

Ages: 2 Days to 2 Days | Sex: All
Age Groups: Child
Study Population: The exploratory nature of this feasibility study dictated to set a realistic target of recruiting 40 preterm infants who are born before 32 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Effect of early Bronchopulmonary dysplasia on the heart right ventricle function. | 20 months
  Establishing sensitive and feasible echo parameters for detecting right ventricle dysfunction associated with early BPD pulmonary vascular changes.

SECONDARY OUTCOMES:
Suitability of eligibility criteria and sample characteristics. | 20 months
  Suitability of eligibility criteria and sample characteristics.
Fidelity to the study procedures. | 20 months
  Fidelity to the study procedures such as recruitment, data collection including echo scans performance at the set time points.
Acquiring relevant data | 20 months
  Recruitment, accrual, and retention rates.

CONTACTS AND LOCATIONS:
Overall Officials: WISAM S MUHSEN, MSc, Study Chair — University of Plymouth; Jos Latour, PhD, Study Director — University of Plymouth; Eirik Nestaas, PhD, Principal Investigator — University of Oslo; Joanne Hosking, PhD, Principal Investigator — University of Plymouth
Locations (1):
- University Hospital Plymouth NHS Trust (UHP), Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appuhn SV, Siebert S, Myti D, Wrede C, Surate Solaligue DE, Perez-Bravo D, Brandenberger C, Schipke J, Morty RE, Grothausmann R, Muhlfeld C. Capillary Changes Precede Disordered Alveolarization in a Mouse Model of Bronchopulmonary Dysplasia. Am J Respir Cell Mol Biol. 2021 Jul;65(1):81-91. doi: 10.1165/rcmb.2021-0004OC. PMID 33784484
- [Background] Alvira CM. Aberrant Pulmonary Vascular Growth and Remodeling in Bronchopulmonary Dysplasia. Front Med (Lausanne). 2016 May 20;3:21. doi: 10.3389/fmed.2016.00021. eCollection 2016. PMID 27243014
- [Background] Ambalavanan N, Mourani P. Pulmonary hypertension in bronchopulmonary dysplasia. Birth Defects Res A Clin Mol Teratol. 2014 Mar;100(3):240-6. doi: 10.1002/bdra.23241. Epub 2014 Mar 10. PMID 24616323
- [Background] Breatnach CR, Levy PT, James AT, Franklin O, El-Khuffash A. Novel Echocardiography Methods in the Functional Assessment of the Newborn Heart. Neonatology. 2016;110(4):248-260. doi: 10.1159/000445779. Epub 2016 Jun 10. PMID 27287615
- [Background] Czernik C, Rhode S, Metze B, Schmalisch G, Buhrer C. Persistently elevated right ventricular index of myocardial performance in preterm infants with incipient bronchopulmonary dysplasia. PLoS One. 2012;7(6):e38352. doi: 10.1371/journal.pone.0038352. Epub 2012 Jun 1. PMID 22675548
- [Background] de Boode WP, Singh Y, Gupta S, Austin T, Bohlin K, Dempsey E, Groves A, Eriksen BH, van Laere D, Molnar Z, Nestaas E, Rogerson S, Schubert U, Tissot C, van der Lee R, van Overmeire B, El-Khuffash A. Recommendations for neonatologist performed echocardiography in Europe: Consensus Statement endorsed by European Society for Paediatric Research (ESPR) and European Society for Neonatology (ESN). Pediatr Res. 2016 Oct;80(4):465-71. doi: 10.1038/pr.2016.126. Epub 2016 Jun 8. No abstract available. PMID 27384404
- [Background] El-Khuffash A, Herbozo C, Jain A, Lapointe A, McNamara PJ. Targeted neonatal echocardiography (TnECHO) service in a Canadian neonatal intensive care unit: a 4-year experience. J Perinatol. 2013 Sep;33(9):687-90. doi: 10.1038/jp.2013.42. Epub 2013 Apr 25. PMID 23619373
- [Background] Erickson CT, Patel MD, Choudhry S, Bisselou KS, Sekarski T, Craft M, Li L, Khuffash AE, Hamvas A, Kutty S, Singh GK, Levy PT. Persistence of right ventricular dysfunction and altered morphometry in asymptomatic preterm Infants through one year of age: Cardiac phenotype of prematurity. Cardiol Young. 2019 Jul;29(7):945-953. doi: 10.1017/S1047951119001161. Epub 2019 Jul 9. PMID 31287038
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Ibrahim J, Bhandari V. The definition of bronchopulmonary dysplasia: an evolving dilemma. Pediatr Res. 2018 Nov;84(5):586-588. doi: 10.1038/s41390-018-0167-9. Epub 2018 Sep 4. PMID 30188504
- [Background] Islam JY, Keller RL, Aschner JL, Hartert TV, Moore PE. Understanding the Short- and Long-Term Respiratory Outcomes of Prematurity and Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2015 Jul 15;192(2):134-56. doi: 10.1164/rccm.201412-2142PP. PMID 26038806
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Khan U, Hjertaas JJ, Greve G, Matre K. Optimal Acquisition Settings for Speckle Tracking Echocardiography-Derived Strains in Infants: An In Vitro Study. Ultrasound Med Biol. 2016 Jul;42(7):1660-70. doi: 10.1016/j.ultrasmedbio.2016.02.015. Epub 2016 Apr 13. PMID 27085385
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077
- [Background] Levy PT, El-Khuffash A, Patel MD, Breatnach CR, James AT, Sanchez AA, Abuchabe C, Rogal SR, Holland MR, McNamara PJ, Jain A, Franklin O, Mertens L, Hamvas A, Singh GK. Maturational Patterns of Systolic Ventricular Deformation Mechanics by Two-Dimensional Speckle-Tracking Echocardiography in Preterm Infants over the First Year of Age. J Am Soc Echocardiogr. 2017 Jul;30(7):685-698.e1. doi: 10.1016/j.echo.2017.03.003. Epub 2017 Apr 19. PMID 28433214
- [Background] Levy PT, Holland MR, Sekarski TJ, Hamvas A, Singh GK. Feasibility and reproducibility of systolic right ventricular strain measurement by speckle-tracking echocardiography in premature infants. J Am Soc Echocardiogr. 2013 Oct;26(10):1201-1213. doi: 10.1016/j.echo.2013.06.005. Epub 2013 Jul 20. PMID 23880052
- [Background] Mertens L, Seri I, Marek J, Arlettaz R, Barker P, McNamara P, Moon-Grady AJ, Coon PD, Noori S, Simpson J, Lai WW; Writing Group of the American Society of Echocardiography (ASE); European Association of Echocardiography (EAE); Association for European Pediatric Cardiologists (AEPC). Targeted neonatal echocardiography in the neonatal intensive care unit: practice guidelines and recommendations for training: Eur J Echocardiogr. 2011 Oct;12(10):715-36. doi: 10.1093/ejechocard/jer181. No abstract available. PMID 21998460
- [Background] Mirza H, Ziegler J, Ford S, Padbury J, Tucker R, Laptook A. Pulmonary hypertension in preterm infants: prevalence and association with bronchopulmonary dysplasia. J Pediatr. 2014 Nov;165(5):909-14.e1. doi: 10.1016/j.jpeds.2014.07.040. Epub 2014 Sep 1. PMID 25189821
- [Background] Mourani PM, Mandell EW, Meier M, Younoszai A, Brinton JT, Wagner BD, Arjaans S, Poindexter BB, Abman SH. Early Pulmonary Vascular Disease in Preterm Infants Is Associated with Late Respiratory Outcomes in Childhood. Am J Respir Crit Care Med. 2019 Apr 15;199(8):1020-1027. doi: 10.1164/rccm.201803-0428OC. PMID 30303395
- [Background] Nestaas E, Schubert U, de Boode WP, El-Khuffash A; European Special Interest Group 'Neonatologist Performed Echocardiography' (NPE). Tissue Doppler velocity imaging and event timings in neonates: a guide to image acquisition, measurement, interpretation, and reference values. Pediatr Res. 2018 Jul;84(Suppl 1):18-29. doi: 10.1038/s41390-018-0079-8. PMID 30072806
- [Background] Sanchez AA, Levy PT, Sekarski TJ, Hamvas A, Holland MR, Singh GK. Effects of frame rate on two-dimensional speckle tracking-derived measurements of myocardial deformation in premature infants. Echocardiography. 2015 May;32(5):839-47. doi: 10.1111/echo.12716. Epub 2014 Aug 11. PMID 25109389
- [Background] Tissot C, Muehlethaler V, Sekarski N. Basics of Functional Echocardiography in Children and Neonates. Front Pediatr. 2017 Dec 1;5:235. doi: 10.3389/fped.2017.00235. eCollection 2017. PMID 29250515
- [Derived] Muhsen WS, Hosking J, Nestaas E, Latour JM. Feasibility of echocardiography and speckle-tracking-derived right ventricular parameters for a prediction model of early bronchopulmonary-dysplasia in preterm infants (REPORT-BPD Study): an observational cohort study. Pilot Feasibility Stud. 2025 Dec 2;12(1):3. doi: 10.1186/s40814-025-01740-3. PMID 41331480
- [Derived] Muhsen WS, Nestaas E, Hosking J, Latour J. Exploring right ventricular function applicability in a prediction model to identify preterm infants with early bronchopulmonary dysplasia (REPORT-BPD study): a mixed-methods observational cohort feasibility study protocol. Pilot Feasibility Stud. 2022 Dec 9;8(1):248. doi: 10.1186/s40814-022-01201-1. PMID 36482482